CLINICAL TRIAL: NCT00722982
Title: Migration Pattern of C-stem AMT Versus Exeter in Total Hip Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Ringerike hospital HF, Hønefoss Norway (Unknown); Ortomedic AS, Lysaker Norway (Unknown); Helse Sor-Ost (Other Government)
Responsible Party: Sponsor
Organization: Oslo University Hospital (Other)
Other Study IDs: C-stem AMT
Record Dates: First submitted 2008-07-25; First posted 2008-07-28 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Coxarthrosis
Keywords: coxarthrosis; hip; RSA; DXA; C-stem AMT; Marathon
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
Hypothesis: Migration of C-Stem AMT is equal to the well documented Exeter prosthesis

In Norway it is annually performed approximately 600 primary and 100 revisions THA. Osteolysis around the prosthesis is one of the major difficulties while performing revision surgery. C-stem is a triple tapered cemented prosthesis designed to increase the stress and strain of proximal femur and thereby decreasing osteolysis. We are planning til include 70 patients and randomize to C-stem AMT or Exeter prosthesis. Both prosthesis will be combined with previously non documented "Marathon" acetabular prosthesis.

The result will be followed clinically and with RSA and DXA. Soft endpoint after 2 years

ELIGIBILITY:
Inclusion Criteria:

* coxarthrosis

Exclusion Criteria:

* age over 80
* major medial condition such as renal failure, chronic obstructive lung disease heart failure etc

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 70 patients admitted to orthopedic clinic Ringerike hospital for coxarthrosis are planned to be included in stydy. The all should agree in a written form to participate in study. They are randomized to be operated THA with Exeter- or C-stem AMT femur prostesis. Marathon acetabular prosthesis will be used for all patients included.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2008-07; Primary Completion 2012-05 (Actual); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Migration of femur- and acetabular prosthesis measured by RSA | 2008-2012

SECONDARY OUTCOMES:
Periprosthetic osteolysis of proximal femur | 2008-2012

CONTACTS AND LOCATIONS:
Overall Officials: Lars Nordsletten, Professor, Study Chair — Ullevaal University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway